CLINICAL TRIAL: NCT04345146
Title: A Prospective, Phase II Study of Bevacizumab Combined With Fractionated Stereotactic Radiotherapy in Patients With 1 to 10 Brain Metastases From Non-small Cell Lung Cancer
Brief Title: Bevacizumab Combined With Fractionated Stereotactic Radiotherapy for 1 to 10 Brain Metastases From NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1053
Record Dates: First submitted 2020-02-22; First posted 2020-04-14 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Bevacizumab; Fractionated stereotactic radiation therapy; Brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FSRT & Bevacizumab (Experimental): Patients will receive Bevacizumab before and after FSRT: daily FSRT(40Gy in 10 fractions or 30Gy in 5 fractions) to the brain metastases with Bevacizumab(7.5mg/kg, q3w, IV)
  Interventions: Combination Product: FSRT combined with Bevacizumab

INTERVENTIONS:
Combination Product: FSRT combined with Bevacizumab — Bevacizumab: Patients will receive Bevacizumab (7.5mg/kg, q3w, IV) before and after FSRT.
  Fractionated stereotactic radiotherapy(FSRT): 40 Gy/10 fractions or 30 Gy/5 fractions for GTV will be delivered to brain metastases.

SUMMARY:
This Phase II randomized study is to determine the efficacy and safety of Bevacizumab combined with fractionated stereotactic radiation therapy(FSRT) in patients with 1 to 10 brain metastases in non-small cell lung cancer by assessing the treatment response, perilesional edema, neurological symptoms and quality of life.

DETAILED DESCRIPTION:
This Phase II randomized study is to determine the efficacy and safety of Bevacizumab combined with fractionated stereotactic radiation therapy(FSRT) in patients with 1 to 10 brain metastases in non-small cell lung cancer by assessing the treatment response, neurological symptoms and quality of life.

Patients will receive Bevacizumab(7.5mg/kg, q3w, i.v.) before and after FSRT(40Gy in 10 fractions or 30Gy in 5 fractions) to the brain metastases. The primary endpoint was intra-cranial progression-free survival (IPFS). Secondary endpoints included overall survival (OS), progression-free survival (PFS), quality of life (QOL) scores, and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years old;
* histologically confirmed NSCLC;
* 1-10 BMs on contrast-enhanced MRI;
* stable extracranial disease status at the time of enrollment;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
* Normal function of organs and bone marrow within 14 days: Total bilirubin 1.5 times or less the upper limits of normal (ULN); AST and ALT 1.5 times or less the ULN; absolute neutrophil count≥ 500 cells/mm3; creatinine clearance rate(CCR) ≥45 mL/min; Platelet count≥50,000 cells/mm3; international normalized ratio(INR) ≤1.5，Prothrombin Time (PT)≤ 1.5 × ULN
* Informed-consent

Exclusion Criteria:

* Intracranial metastases needed surgical decompression
* Patients with contraindications for MRI
* Previous radiotherapy or excision for intracranial metastases
* The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava)
* A cavity over 2cm in diameter of primary tumor or metastasis
* Bleeding tendency or coagulation disorder
* Hemoptysis (1/2 teaspoon blood/day) happened within 1 month
* The use of full-dose anticoagulation within the past 1 month
* Severe vascular disease occurred within 6 months
* Gastrointestinal fistula, perforation or abdominal abscess occurred within 6 months
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg)
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours
* Urine protein 3-4+, or 24h urine protein quantitative >1g
* Severe uncontrolled disease
* Uncontrollable seizure or psychotic patients without self-control ability
* Women in pregnancy, lactation period
* Other not suitable conditions determined by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Intracranial progression-free survival | 1 year
  IPFS was calculated from the completion of radiotherapy until the first occurrence of either intracranial progression or death.

SECONDARY OUTCOMES:
overall survival (OS) | 1 year
progression-free survival (PFS) | 1 year
Rate of participants with perilesional edema of brain metastases evaluated by T2-weighted MRI | 1 year
Quality of life evaluated by EORTC quality of life questionnaire | 6 months
  Quality of life evaluated by EORTC quality of life questionnaire(QLQ-C30 and QLQ-BN20)
Rate of patients with treatment-related adverse events evaluated by CTCAE v5.0 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Shaw MG, Ball DL. Treatment of brain metastases in lung cancer: strategies to avoid/reduce late complications of whole brain radiation therapy. Curr Treat Options Oncol. 2013 Dec;14(4):553-67. doi: 10.1007/s11864-013-0258-0. PMID 24048959
- [Background] Yuan X, Liu WJ, Li B, Shen ZT, Shen JS, Zhu XX. A Bayesian network meta-analysis of whole brain radiotherapy and stereotactic radiotherapy for brain metastasis. Medicine (Baltimore). 2017 Aug;96(34):e7698. doi: 10.1097/MD.0000000000007698. PMID 28834873
- [Background] Magnuson WJ, Lester-Coll NH, Wu AJ, Yang TJ, Lockney NA, Gerber NK, Beal K, Amini A, Patil T, Kavanagh BD, Camidge DR, Braunstein SE, Boreta LC, Balasubramanian SK, Ahluwalia MS, Rana NG, Attia A, Gettinger SN, Contessa JN, Yu JB, Chiang VL. Management of Brain Metastases in Tyrosine Kinase Inhibitor-Naive Epidermal Growth Factor Receptor-Mutant Non-Small-Cell Lung Cancer: A Retrospective Multi-Institutional Analysis. J Clin Oncol. 2017 Apr 1;35(10):1070-1077. doi: 10.1200/JCO.2016.69.7144. Epub 2017 Jan 23. PMID 28113019
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Background] Aoyama H, Tago M, Kato N, Toyoda T, Kenjyo M, Hirota S, Shioura H, Inomata T, Kunieda E, Hayakawa K, Nakagawa K, Kobashi G, Shirato H. Neurocognitive function of patients with brain metastasis who received either whole brain radiotherapy plus stereotactic radiosurgery or radiosurgery alone. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1388-95. doi: 10.1016/j.ijrobp.2007.03.048. PMID 17674975
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Serizawa T, Yamamoto M, Higuchi Y, Sato Y, Shuto T, Akabane A, Jokura H, Yomo S, Nagano O, Kawagishi J, Yamanaka K. Local tumor progression treated with Gamma Knife radiosurgery: differences between patients with 2-4 versus 5-10 brain metastases based on an update of a multi-institutional prospective observational study (JLGK0901). J Neurosurg. 2019 Apr 26;132(5):1480-1489. doi: 10.3171/2019.1.JNS183085. Print 2020 May 1. PMID 31026833
- [Background] Rades D, Janssen S, Dziggel L, Blanck O, Bajrovic A, Veninga T, Schild SE. A matched-pair study comparing whole-brain irradiation alone to radiosurgery or fractionated stereotactic radiotherapy alone in patients irradiated for up to three brain metastases. BMC Cancer. 2017 Jan 6;17(1):30. doi: 10.1186/s12885-016-2989-3. PMID 28061768
- [Background] Manning MA, Cardinale RM, Benedict SH, Kavanagh BD, Zwicker RD, Amir C, Broaddus WC. Hypofractionated stereotactic radiotherapy as an alternative to radiosurgery for the treatment of patients with brain metastases. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):603-8. doi: 10.1016/s0360-3016(00)00475-2. PMID 10837942
- [Background] Baliga S, Garg MK, Fox J, Kalnicki S, Lasala PA, Welch MR, Tome WA, Ohri N. Fractionated stereotactic radiation therapy for brain metastases: a systematic review with tumour control probability modelling. Br J Radiol. 2017 Feb;90(1070):20160666. doi: 10.1259/bjr.20160666. Epub 2016 Dec 12. PMID 27936894
- [Background] Mekhail T, Sombeck M, Sollaccio R. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. Curr Oncol Rep. 2011 Aug;13(4):255-8. doi: 10.1007/s11912-011-0180-1. No abstract available. PMID 21584645
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Barrett OC, McDonald AM, Thompson JW, Bredel M, McGwin G, Riley KO, Fiveash JB. Distant brain recurrence in patients with five or more newly diagnosed brain metastases treated with focal stereotactic radiotherapy alone. J Radiosurg SBRT. 2017;4(4):255-263. PMID 28626600
- [Background] Socinski MA, Langer CJ, Huang JE, Kolb MM, Compton P, Wang L, Akerley W. Safety of bevacizumab in patients with non-small-cell lung cancer and brain metastases. J Clin Oncol. 2009 Nov 1;27(31):5255-61. doi: 10.1200/JCO.2009.22.0616. Epub 2009 Sep 8. PMID 19738122
- [Background] Zustovich F, Ferro A, Lombardi G, Zagonel V, Fiduccia P, Farina P. Bevacizumab as front-line treatment of brain metastases from solid tumors: a case series. Anticancer Res. 2013 Sep;33(9):4061-5. PMID 24023350
- [Background] Jiang T, Zhang Y, Li X, Zhao C, Chen X, Su C, Ren S, Yang N, Zhou C. EGFR-TKIs plus bevacizumab demonstrated survival benefit than EGFR-TKIs alone in patients with EGFR-mutant NSCLC and multiple brain metastases. Eur J Cancer. 2019 Nov;121:98-108. doi: 10.1016/j.ejca.2019.08.021. Epub 2019 Sep 27. PMID 31569068
- [Background] Boothe D, Young R, Yamada Y, Prager A, Chan T, Beal K. Bevacizumab as a treatment for radiation necrosis of brain metastases post stereotactic radiosurgery. Neuro Oncol. 2013 Sep;15(9):1257-63. doi: 10.1093/neuonc/not085. Epub 2013 Jun 27. PMID 23814264
- [Background] Yomo S, Hayashi M. Salvage stereotactic radiosurgery with adjuvant use of bevacizumab for heavily treated recurrent brain metastases: a preliminary report. J Neurooncol. 2016 Mar;127(1):119-26. doi: 10.1007/s11060-015-2019-3. Epub 2015 Nov 30. PMID 26619997
- [Background] Xiangying M, Rugang Z, Lijuan D, Yaowei Z, Bing S, Junliang W, Dan L, Shikai W. Low-dose bevacizumab as an effective pre-treatment for peri-tumoral brain edema prior to CyberKnife radiosurgery: A case report. Cancer Biol Ther. 2018 Jun 3;19(6):461-464. doi: 10.1080/15384047.2018.1433499. Epub 2018 Mar 21. PMID 29420112
- [Background] Levy C, Allouache D, Lacroix J, Dugue AE, Supiot S, Campone M, Mahe M, Kichou S, Leheurteur M, Hanzen C, Dieras V, Kirova Y, Campana F, Le Rhun E, Gras L, Bachelot T, Sunyach MP, Hrab I, Geffrelot J, Gunzer K, Constans JM, Grellard JM, Clarisse B, Paoletti X. REBECA: a phase I study of bevacizumab and whole-brain radiation therapy for the treatment of brain metastasis from solid tumours. Ann Oncol. 2015 Nov;26(11):2359. doi: 10.1093/annonc/mdv386. No abstract available. PMID 26504187
- [Background] Clarke J, Neil E, Terziev R, Gutin P, Barani I, Kaley T, Lassman AB, Chan TA, Yamada J, DeAngelis L, Ballangrud A, Young R, Panageas KS, Beal K, Omuro A. Multicenter, Phase 1, Dose Escalation Study of Hypofractionated Stereotactic Radiation Therapy With Bevacizumab for Recurrent Glioblastoma and Anaplastic Astrocytoma. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):797-804. doi: 10.1016/j.ijrobp.2017.06.2466. Epub 2017 Jun 30. PMID 28870792
- [Background] Eisele SC, Wen PY, Lee EQ. Assessment of Brain Tumor Response: RANO and Its Offspring. Curr Treat Options Oncol. 2016 Jul;17(7):35. doi: 10.1007/s11864-016-0413-5. PMID 27262709
- [Derived] Zhou R, Zheng S, Wang D, Dong F, Zhang H, Zhang T, Luo Q, Liu B, Liu H, Zhang J, Liu F, Wang B, Chen L, Mou Y, Peng K, Qiu B, Liu H. Efficacy and safety of combining bevacizumab and fractionated stereotactic radiotherapy for extensive brain metastases in patients with non-small cell lung cancer: a prospective phase II study (GASTO-1053). Cancer Commun (Lond). 2025 Dec;45(12):1739-1754. doi: 10.1002/cac2.70078. Epub 2025 Nov 14. PMID 41235462